CLINICAL TRIAL: NCT04236843
Title: Faecal Microbiota Transplantation (FMT) in Patients With Irritable Bowel Syndrome (IBS): Optimizing the Treatment and Its Mechanism(s) of Action
Brief Title: Faecal Microbiota Transplantation (FMT) in Patients With IBSmechanism(s) of Action
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helse Fonna (Other)
Collaborators: University of Bergen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Helse Fonna
Record Dates: First submitted 2020-01-15; First posted 2020-01-22 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Irritable Bowel Syndrome
Keywords: Fecal microbiota transplantation; Intestinal microbiota; Donor; Dysbiosis; Abdominal symptom; Fatigue; Quality of life
MeSH Terms: conditions — Irritable Bowel Syndrome; Dysbiosis; Fatigue | interventions — Defecation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Smal intestine once (Active Comparator): 90-g fecal transplant given into the small intestine once.
  Interventions: Dietary Supplement: Feces
- Small intestine twice (Active Comparator): 90-g fecal transplant given into the small intestine twice with 1 week interval.
  Interventions: Dietary Supplement: Feces
- Large intestine once (Active Comparator): 90-g fecal transplant given into the large intestine once.
  Interventions: Dietary Supplement: Feces

INTERVENTIONS:
Dietary Supplement: Feces — Feces from healthy donor

SUMMARY:
Two hundrad patients are randomized to either 90 g transplant, 90 g transplant twice with 1week interval into the distal small intestine via working channel of a gastroscope, or to 90 g transplant into the coecum of the colon via working channel of a colonoscope. The patients shall complete 5 questionnaires measuring symptoms, fatigue and quality of life and collect a feces sample at the baseline, and at 3, 6 and 12 months after FMT. Dysbiosis and fecal bacterial are determined by using 16S rRNA gene.

DETAILED DESCRIPTION:
Patients Two hundrad patients who fulfil Rome IV criteria for irritable bowel syndrome (IBS) shall be included in the study. All the IBS subtypes shall be included.

Donor Investigators are going to use the same super-donor they used in their previous randomised double-blind, placebo-controlled study. The donor is athletic Caucasian man aging 36 years. He is non-smoker and is completely healthy without any medication and with a BMI of 23.5. He is not relative to any of the patients in the trial. He was borne by vaginal delivery and breastfeed. He was treated 3 times with antibiotics during his life. He trains 5 times weekly an hour each time. He took regularly dietary supplements rich in proteins, vitamins, fibres and minerals that made his diet richer than average in these substances. He was screened according to the guidelines for donors for FMT. Before he was accepted as a donor the microbiota was analysed in a faecal sample using GA-map Dysbiosis test. The analysis revealed a dysbiosis index (DI)= 1, indicating normobiosysis. In addition, he had excess of bacteria belonging to the Firmicutes. His faeces shall be tested every third moth during the trial.

Protocol

The patients are randomized to either 90 g transplant, 90 g transplant twice with 1week interval into the distal small intestine, or to 90 g transplant into the coecum of the colon. The patients shall complete 5 questionnaires and deliver fecal samples at the baseline, and at 3 , 6 , and 12 months after FMT.

Faeces collection, preparation and administration Faeces from both the donor and patients shall be collected and stored at - 80•. Frozen faeces shall be thawed and each 30 g is dissolved in 30 mL of 0.9% sterile saline. The dissolved stool administrated to the patients, after overnight fast, through working channel of gastroduodeno-scope in pars descendent duodenum distal to the papilla of Vater or to the coecum through working channel of a colonoscope.

Analysis Questionnaires

1. IBS symptom severity Scale (IBS-SSS).
2. Birmingham Symptom scale.
3. IBS-quality of life (IBSQo) Questionnaire.
4. Short form of Nepean Dyspepsia Index (SF-NDI).
5. Fatigue Assessment Scale (FAS).

Microbiome analysis Gut microbiota analysis is performed using the Genetic analysis-mapTM Dysbiosis test (Genetic Analysis AS, Oslo, Norway) by algorithmically assessing faecal bacterial abundance and profile (dysbiosis index, DI), and potential deviation in the microbiome from normobiosis. GA-map test is based on faecal homogenization, mechanical bacterial cell disruption and automated total bacterial genomic DNA extraction using magnetic beads. DI is based on 54 DNA probes targeting more than 300 bacterial strains based on their 16S rRNA sequence in seven variable regions (V3-V9). Twenty-six bacteria probes are species specific, 19 detect bacteria on genus level, and 9 probes detect bacteria at higher taxonomic levels. Probe labelling is by single nucleotide extension and hybridization to complementary probes coupled to magnetic beads, and signal detection by using BioCode 1000A 128-Plex Analyser (Applied BioCode, Santa Fe Springs, CA, USA). A DI above 2 shows a microbiota profile that differs from that of the normobiotic reference collection (DI 1-2: non-dysbiosis, DI: moderate, DI 4-5: severe dysbiosis).

ELIGIBILITY:
Inclusion Criteria:

1. Patients who fulfil Rome IV criteria for the diagnosis of IBS.
2. Patients were investigated to exclude other gastrointestinal organic cause(s).
3. Moderate-to-severe IBS symptoms, as indicated by a score of ≥175 on the IBS Severity Scoring System (IBS-SSS).

Exclusion Criteria:

1. Pregnant or lactating women.
2. The use of antibiotics or probiotics within 1 month prior to FMT.
3. Immunocompromised patients defined as those treated by immune- suppressive medications.
4. Patients with co-morbidity such as kidney failure or chronic heart disease.
5. System disease such as diabetes.
6. Patients with serious psychiatric disorders or drug abuse.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Actual)
Dates: Start 2020-02-03 (Actual); Primary Completion 2022-03-25 (Actual); Study Completion 2022-03-25 (Actual)

PRIMARY OUTCOMES:
Change in IBS-SSS total score | 12 months after FMT
  Irritable bowel syndrome-symptom severity score (IBS-SSS) is a visual analogue scale questionnaire with a maximum score of 500 points. A decrease in total score by ≥50 points is considered as a response.

SECONDARY OUTCOMES:
Change in the Dysbiosis index | 12 months after FMT
  Dysbiosis index (DI) is a 5 -scale index. A DI above 2 shows a microbiota profile that differs from that of the normobiotic reference collection (DI 1-2: non-dysbiosis, DI 3: moderate, DI 4-5: severe dysbiosis)

CONTACTS AND LOCATIONS:
Overall Officials: Magdy El-Salhy, MD,PhD, Study Chair — Helse Fonna
Locations (1):
- Helse Fonna, Haugesund, Norway

REFERENCES:
- [Derived] El-Salhy M, Gilja OH, Hatlebakk JG. Factors underlying the long-term efficacy of faecal microbiota transplantation for patients with irritable bowel syndrome. Microbes Infect. 2024 Nov-Dec;26(8):105372. doi: 10.1016/j.micinf.2024.105372. Epub 2024 Jun 4. PMID 38843950
- [Derived] El-Salhy M, Hatlebakk JG. Factors Underlying the Difference in Response to Fecal Microbiota Transplantation Between IBS Patients with Severe and Moderate Symptoms. Dig Dis Sci. 2024 Apr;69(4):1336-1344. doi: 10.1007/s10620-024-08369-x. Epub 2024 Mar 6. PMID 38446309
- [Derived] El-Salhy M, Gilja OH, Hatlebakk JG. Increasing the transplant dose and repeating faecal microbiota transplantation results in the responses of male patients with IBS reaching those of females. Scand J Gastroenterol. 2024 Apr;59(4):391-400. doi: 10.1080/00365521.2023.2292479. Epub 2023 Dec 12. PMID 38084725
- [Derived] El-Salhy M, Gilja OH, Hatlebakk JG. Factors affecting the outcome of fecal microbiota transplantation for patients with irritable bowel syndrome. Neurogastroenterol Motil. 2024 Jan;36(1):e14641. doi: 10.1111/nmo.14641. Epub 2023 Jul 10. PMID 37427566